CLINICAL TRIAL: NCT04718805
Title: A Single-dose, Open-label, Randomized, Crossover Pivotal Bioequivalence Study in Healthy Participants to Assess the Bioequivalence of Darunavir 675 mg in the Presence of 150 mg Cobicistat When Administered as a Fixed Dose Combination (Darunavir/Cobicistat) Compared to the Co-administration of the Separate Agents (Darunavir and Cobicistat) Under Fed Conditions
Brief Title: A Study of Darunavir in the Presence of Cobicistat When Administered as a Fixed Dose Combination Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CR108955; TMC114IFD1004 (Other: Janssen Research & Development, LLC); 2020-003397-43 (EudraCT Number)
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Darunavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment A (Experimental): Participants will receive Treatment A (a single dose of darunavir [DRV]/cobicistat [COBI] as one fixed dose combination [FDC] tablet under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence AB or BA). A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir; Drug: Cobicistat; Drug: Darunavir/Cobicistat FDC
- Treatment B (Active Comparator): Participants will receive Treatment B (a single dose of DRV/COBI as separate tablets under fed condition on Day 1) as per assigned treatment sequence (Treatment sequence BA or AB). A washout period of at least 7 days will be maintained between each treatment period.
  Interventions: Drug: Darunavir; Drug: Cobicistat

INTERVENTIONS:
Drug: Darunavir — Participants will receive a single dose of Darunavir tablets orally as per assigned treatment sequence.
  Other Names: TMC114
Drug: Cobicistat — Participant will receive a single dose of Cobicistat tablets orally as per assigned treatment sequence.
  Other Names: JNJ-48763364
Drug: Darunavir/Cobicistat FDC — Participants will receive a single dose of darunavir and cobicistat FDC tablets orally as per assigned treatment sequence.
  Arms: Treatment A

SUMMARY:
The purpose of this study is to evaluate the single-dose Pharmacokinetic (PK) and bioequivalence of darunavir (DRV) in the presence of cobicistat (COBI) when administered as a scored fixed dose combination (FDC) tablet (DRV/COBI) compared to the co-administration as the separate available tablet formulations (DRV and COBI), under fed conditions in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 30.0 kilograms per meter square (kg/m^2) inclusive, and body weight not less than 50.0 kg
* Must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* Must be healthy on the basis of clinical laboratory tests performed at screening
* Non-postmenopausal women must have a negative highly sensitive serum beta-human chorionic gonadotropin (beta- hCG) 4 days or less before dosing of the first treatment period
* A woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 90 days after receiving the last dose of study drug
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies
* Must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* During the study and for a minimum of at least 90 days after receiving the last dose of study drug, a male participant: must wear a condom when engaging in any activity that allows for passage of ejaculate to another person (male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak), must agree not to donate sperm for the purpose of reproduction

Exclusion Criteria:

* Has a history of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Has received an investigational drug or used an investigational medical device within 60 days before the first administration of the study drug
* Has a history of hepatitis A antibody immunoglobulin M (IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for hepatitis A antibody IgM, HBsAg or anti-HCV at screening
* Has previously participated in more than 3 single-dose trials or a multiple-dose trial with darunavir (DRV) and/or cobicistat (COBI)
* Has had any contact with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positive or Coronavirus Disease 2019 (COVID-19) patients within the last 2 weeks prior to admission to the clinical research center
* Is a woman who is pregnant, breast-feeding, or planning to become pregnant during the study or within 90 days after the last dose of study drug, or a woman of childbearing potential who is unwilling to use acceptable methods of contraception
* Has a history of human immunodeficiency virus type 1 or type 2 (HIV-1 or HIV-2) antibody positive, or tests positive for HIV at screening
* Positive test for SARS-CoV-2 test participants within the last 2 weeks prior to admission or during the study
* Is a man who plans to father a child while enrolled in the study or within 90 days after the last dose of study drug, or who is unwilling to use acceptable methods of contraception

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Analyte Concentration (Cmax) of Darunavir (DRV) | Predose, up to 72 hours post dose (up to Day 4)
  Cmax is defined as the maximum observed analyte concentration of DRV.
Area Under the Analyte Concentration-time Curve from time Zero to Last Quantifiable time (AUC[0-last]) of DRV | Predose, up to 72 hours post dose (up to Day 4)
  AUC(0-last) is the area under the analyte concentration-time curve from time zero to the time of the last measurable (non-below quantification limit [non-BQL]) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of DRV | Predose, up to 72 hours post dose (up to Day 4)
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z), wherein AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, Clast is the last observed measurable (non-BQL) concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 6 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Cmax of Cobicistat (COBI) | Predose, up to 72 hours post dose (up to Day 4)
  Cmax is defined as the maximum observed analyte concentration of COBI.
Area Under the Analyte Concentration-time Curve from time Zero to Last Quantifiable time (AUC[0-last]) of COBI | Predose, up to 72 hours post dose (up to Day 4)
  AUC(0-last) is the area under the analyte concentration-time curve from time zero to the time of the last measurable (non-BQL) concentration, calculated by linear-linear trapezoidal summation.
Area Under the Analyte Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of COBI | Predose, up to 72 hours post dose (up to Day 4)
  AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(last)/lambda(z), wherein AUC(0-last) is area under the analyte concentration-time curve from time zero to last quantifiable time, Clast is the last observed measurable (non-BQL) concentration, and lambda(z) is elimination rate constant.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- SGS Clinical Pharmacology Unit (located in ZNA Stuivenberg), Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency